CLINICAL TRIAL: NCT06602583
Title: Radiation Exposure in Diagnostic Angiography With and Without a New Low Dose Exposure Protocol -Radiation Exposure Reduction Study
Brief Title: To Determine the Difference in the Radiation Exposure, With Low Dose Protocols for Angiography
Acronym: RADRED
Status: Not yet recruiting | Type: Observational
Sponsor: Dr Bharat Singh Sambyal (Other Government)
Responsible Party: Sponsor-Investigator, Dr Bharat Singh Sambyal, Principal Investigator, Institute of Naval Medicine, Indian Naval Hospital Ship (INHS) Asvini
Organization: Institute of Naval Medicine, Indian Naval Hospital Ship (INHS) Asvini (Other Government)
Other Study IDs: REF/2024/09/092182
Record Dates: First submitted 2024-09-17; First posted 2024-09-19 (Actual); Last update posted 2024-09-20 (Actual); Status verified 2024-09

CONDITIONS: Coronary Arterial Disease (CAD)
Keywords: coronary angiography; coronary artery disease; radiation exposure; DAP; KAP
MeSH Terms: conditions — Coronary Artery Disease | interventions — Coronary Angiography; Angiography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- A study arm 1: baseline comparative arm of patients having already undergone angiography and fitting the inclusion criteria. The radiation exposure of this group would be collected from database of already done studies in the months prior to the initiation of the study (so as to prevent observer bias which may happen once the interventional cardiologist knows his inclusion in study, and may use a shorter or longer cine runs, thus influencing the outcomes). This would best represent the real-world data set, according to the routinely followed standard dose/ older low dose protocol.
  Interventions: Diagnostic Test: Standard Dose Coronary angiography
- A study arm 2: a comparative arm where the patients being once eligible for the study; would undergo angiography using the new low dose protocol. A total of 5 to 8 different views (orthogonal) would be taken (2 for RCA and 4 to 6 for LAD/LCX)
  Interventions: Diagnostic Test: New low dose angiography

INTERVENTIONS:
Diagnostic Test: Standard Dose Coronary angiography — The radiation exposure of this group would be collected from database of already done studies in the months prior to the initiation of the study (so as to prevent observer bias which may happen once the interventional cardiologist knows his inclusion in study, and may use a shorter or longer cine runs, thus influencing the outcomes). This would best represent the real-world data set, according to the routinely followed standard dose/ older low dose protocol.
  Other Names: Standard Dose Angiography
  Groups: A study arm 1
Diagnostic Test: New low dose angiography — a comparative arm where the patients being once eligible for the study; would undergo angiography using the new low dose protocol.
  Groups: A study arm 2

SUMMARY:
1. The patients suspected coronary artery disease or those needing an angiography as per the inclusion criteria would be included after a 2d echocardiography and treadmill test/ stress myocardial stress imaging (if indicated) after a written and informed consent.
2. Anthropometric and lab paraments would be recorded.
3. Study will have 2 arms. I. A study arm 1 - baseline comparative arm of patients having undergone angiography with standard dose/ old low dose angiography.

   II. A study arm 2 - a comparative arm where the patients being once eligible for the study; would undergo angiography using the new low dose protocol.
4. Post completion of the sample size the data of each angiographic view would be noted in both the study arms

DETAILED DESCRIPTION:
INTRODUCTION

The increasing prevalence of cardiovascular diseases has led to a surge in the use of diagnostic angiography procedures. While these procedures are crucial for diagnosing and treating heart conditions, they also involve significant exposure to ionizing radiation. Excessive radiation exposure can pose serious health risks, including an increased risk of cancer and other adverse effects.

The RADRED study aims to address the critical issue of radiation exposure in cardiology catheterization labs. By comparing the radiation dose received by patients undergoing diagnostic angiography with and without a new low dose exposure protocol, the study seeks to evaluate the effectiveness of this protocol in reducing radiation exposure.

Several factors contribute to the need for such research. Firstly, the growing number of patients undergoing diagnostic angiography, particularly elderly individuals and those with multiple comorbidities, increases the cumulative radiation exposure to the population. Secondly, advancements in imaging technology have led to more complex procedures, often requiring longer fluoroscopy times, which can result in higher radiation doses. Finally, there is a growing awareness of the potential long-term health consequences of radiation exposure, particularly for vulnerable populations.

The RADRED study has the potential to make a significant contribution to the field of cardiology by demonstrating the feasibility and benefits of implementing a low dose exposure protocol in catheterization labs. By reducing radiation exposure, this protocol can help to protect the health of patients and healthcare providers, while also improving the overall efficiency and cost-effectiveness of diagnostic angiography procedures AIM To study determine the difference in the radiation exposure in diagnostic angiography with and without a new low dose exposure protocol

OBJECTIVES Primary objective To determine the difference in the radiation exposure levels received by patients undergoing diagnostic angiography with and without the new low dose exposure protocol.

Secondary objectives

1. To evaluate the diagnostic image quality obtained with the new low dose exposure protocol compared to the standard protocol.
2. To assess any potential limitations associated with the new low dose exposure protocol.

STUDY DESIGN:

Observational analytical cohort study

PARTICIPANTS:

Inclusion criteria:

Adult patients who qualify for a need of diagnostic angiography and are finally found to have normal epicardial coronaries, e.g.:

* Pre aortic or mitral valve replacement angiography
* TMT positive for inducible ischemia
* SPECT MPI positive patients
* Cradiologically symptomatic patients with ECG abnormalities, who cannot be subjected to stress test
* High risk pre transplant patients

Exclusion criteria:

* Those who are unwilling for study
* Patients who come with STEMI or NSTEMI

STUDY METHOD:

1. The patients suspected coronary artery disease or those needing an angiography as per the inclusion criteria would be included after a 2d echocardiography and treadmill test/ stress myocardial stress imaging (if indicated) after a written and informed consent.
2. Anthropometric and lab paraments would be recorded.
3. Study will have 2 arms. I. A study arm 1 - baseline comparative arm of patients having undergone angiography with standard dose/ old low dose angiography.

   II. A study arm 2 - a comparative arm where the patients being once eligible for the study; would undergo angiography using the new low dose protocol.
4. Post completion of the sample size the data of each angiographic view would be noted in both the study arms

PERIOD OF STUDY: till completion of sample in study arm 2 (each successive patient would be enrolled - cluster sample)

PATIENT CONSENT:

Appropriate approval will be obtained from IEC of the institute.

STATISTCAL ANALYSIS Data will be compiled in an excel sheet for all the variables of interest and presented in the form of tables and graphs as appropriate.

Measures of central tendency (mean or median) would be calculated for all quantitative variables along with measures of dispersion (standard deviation or interquartile range). Qualitative or categorical variables will be described as frequencies and proportions. The investigators will use a t-test for independent samples to compare the means of radiation exposure All the statistical analysis will be carried out using Statistical Package for Social Sciences (SPSS Inc., Chicago, IL, version 22.0 for Windows) at 5% level of significance i.e., p≤0.05 will be considered significant

ETHICAL JUSTIFICATION This study aims to evaluate the efficacy of a new low-dose radiation protocol for diagnostic angiography in cardiology Cath labs. By comparing patient radiation exposure with and without the protocol, the study seeks to reduce the cumulative radiation burden on patients, especially those at higher risk due to age or underlying health conditions. The increasing frequency of diagnostic angiography, coupled with advancements in imaging technology leading to more complex procedures, has resulted in a growing concern about the potential long-term health risks associated with radiation exposure. This study addresses this critical issue by exploring the effectiveness of a new protocol designed to minimize radiation dose during these procedures

. As, such low dose protocol has never been used earlier, there is a need for evaluating the same as to set new standards and protocols

The patients involved in the research project will be informed of the methods, anticipated benefits and potential risks of the study and the discomfort it may cause and the remedies thereof.

Written informed consent will be obtained. Every precaution will be taken to respect the privacy and confidentiality of the patient.

The parent has right to abstain from the study or to withdraw consent to participate at any time of the study without reprisal.

Due care and caution will be taken at all stages to ensure that the patient is put to minimum risk or suffer from irreversible side effects and probably benefit from study

DISCLOSURES/ CONFLICT OF INTEREST: NIL

ELIGIBILITY:
Inclusion Criteria:

Adult patients who qualify for a need of diagnostic angiography and are finally found to have normal epicardial coronaries, e.g.:

* Pre aortic or mitral valve replacement angiography
* TMT positive for inducible ischemia
* SPECT MPI positive patients
* Cradiologically symptomatic patients with ECG abnormalities, who cannot be subjected to stress test
* High risk pre transplant patients

Exclusion Criteria:

* Those who are unwilling for study
* Patients who come with STEMI or NSTEMI

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing diagnostic angiography (age ≥18 years) will be included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2024-10-01 (Estimated); Primary Completion 2025-02-28 (Estimated); Study Completion 2025-04-30 (Estimated)

PRIMARY OUTCOMES:
To determine the difference in the radiation exposure levels received by patients undergoing diagnostic angiography with and without the new low dose exposure protocol | Through study completion, and average of 06 monhts
  Study aims to address the critical issue of radiation exposure in cardiology catheterization labs. By comparing the radiation dose received by patients undergoing diagnostic angiography with and without a new low dose exposure protocol, the study seeks to evaluate the effectiveness of this protocol in reducing radiation exposure.

CONTACTS AND LOCATIONS:
Overall Officials: Dr Bharat S Sambyal, DM Card, Principal Investigator — INHS Asvini; Dr R Anathakrishnan, DM Card, Study Director — INHS Asvini
Locations (1):
- INHS Asvini, Mumbai, Maharashtra, India

IPD SHARING:
Plan to Share IPD: Undecided
Currently there is no plan to share the IPD data due to government hospital data sharing restrictions. though anonymous data can be shared with a fellow researcher if a combined study is planned

REFERENCES:
- [Background] Picano E. Sustainability of medical imaging. BMJ. 2004 Mar 6;328(7439):578-80. doi: 10.1136/bmj.328.7439.578. PMID 15001510
- [Background] Padovani R, Le Heron J, Cruz-Suarez R, Duran A, Lefaure C, Miller DL, Sim HK, Vano E, Rehani M, Czarwinski R. International project on individual monitoring and radiation exposure levels in interventional cardiology. Radiat Prot Dosimetry. 2011 Mar;144(1-4):437-41. doi: 10.1093/rpd/ncq326. Epub 2010 Nov 3. PMID 21051431
- [Background] Stocker TJ, Abdel-Wahab M, Mollmann H, Deseive S, Massberg S, Hausleiter J. Radiation Dose in Diagnostic Cardiac Catheterization: Results From the PROTECTION VII Study. JACC Cardiovasc Interv. 2021 Sep 13;14(17):1958-1960. doi: 10.1016/j.jcin.2021.07.023. No abstract available. PMID 34503751
- [Background] Tong J, Hei TK. Aging and age-related health effects of ionizing radiation. Radiat Med Prot [Internet]. 2020 Mar 1 [cited 2024 Sep 10];1(1):15-23. Available from: https://www.sciencedirect.com/science/article/pii/S2666555720300058
- [Background] Kar S, Teleb M, Albaghdadi A, Ibrahim A, Mukherjee D. Efficacy of Low-Dose Compared With Standard-Dose Radiation for Cardiac Catheterization and Intervention (KAR RAD Study). J Invasive Cardiol. 2019 Jun;31(6):187-194. doi: 10.25270/jic/18.00332. Epub 2019 Mar 15. PMID 30865914
- See also: Radiation Units and Conversion Factors - Radiation Emergency Medical Management [Internet]. [cited 2024 Sep 10]. — https://remm.hhs.gov/radmeasurement.htm